CLINICAL TRIAL: NCT03700411
Title: Influence of Peri-operative Opioid Analgesia on Circulating Tumor Cells in Patients Undergoing Open Colorectal Cancer Surgery - Multi-center, Randomized Clinical Trial
Brief Title: Influence of Opioid Analgesia on Circulating Tumor Cells in Open Colorectal Cancer Surgery
Acronym: POACC-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other); Tomas Bata Hospital, Czech Republic (Other); University Hospital Ostrava (Other); Hospital Novy Jicin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POACC-1
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Circulating Tumor Cell
Keywords: Perioperative analgesia; Colorectal Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating | interventions — Morphine; Pirinitramide; Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morphine (Active Comparator): Morphine-based perioperative analgesia
  Interventions: Drug: Morphine
- Piritramid (Active Comparator): Piritramid-based perioperative analgesia
  Interventions: Drug: Piritramid
- Epidural (Active Comparator): Perioperative epidural analgesia containing an opioid
  Interventions: Drug: Epidural

INTERVENTIONS:
Drug: Morphine — Morphine intravenous
  Arms: Morphine
Drug: Piritramid — Piritramid intravenous
  Arms: Piritramid
Drug: Epidural — Perioperative epidural analgesia
  Arms: Epidural

SUMMARY:
To compare the effects of three types of perioperative analgesia on the number of circulating tumor cells following radical colorectal cancer surgery. To find correlations with other perioperative factors and clinical/pathological disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing open radical surgery for colorectal cancer
* age over 18 years
* signed informed consent

Exclusion Criteria:

* intolerance of the study drugs
* history of CRC surgery
* neoadjuvant therapy
* contraindications to epidural analgesia
* other malignancy not in permanent remission
* chronic opioid medication or opioid administration within 7 days preoperatively
* immunosuppressive or corticosteroid therapy
* surgery within 30 days preoperatively (except minor)
* chronic or acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Change in number of circulating tumor cells prior to surgery to 2 - 4 weeks after surgery | 1 - 3 days before surgery to 4 weeks after surgery
  Baseline number of circulating tumor cells will be recorded prior to surgery in a venous blood sample. Number of circulating tumor cells will be measured 2 - 4 weeks after surgery in a venous blood sample. These two values will be compared.

SECONDARY OUTCOMES:
Pain assessment | 3 days postoperatively
  Pain intensity assessed using Numerical Rating Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD PhD, Principal Investigator — Institute of Molecular and Translational Medicine, Palacky University, Olomouc
Locations (3):
- Czechia (3):
  - T. Bata Regional Hospital Zlin, Zlin, South Moravian
  - University Hospital Ostrava, Ostrava
  - General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berta E, Srovnal J, Dytrych P, Bruthans J, Ulrichova J, Prasil P, Vecera L, Gabrhelik T, Tolmaci B, Dusa J, Maca J, Mazancova M, Haiduk F, Kutej M, Ihnat P, Michalek P, Hajduch M. Influence of opioid analgesia type on circulating tumor cells in open colorectal cancer surgery (POACC-1): study protocol for a prospective randomized multicenter controlled trial. BMC Anesthesiol. 2023 Feb 28;23(1):64. doi: 10.1186/s12871-023-02007-1. PMID 36855089